CLINICAL TRIAL: NCT01510886
Title: Assessment of MDD Management Strategies in Andalusia: A Sub-analysis of the PismaEP Study
Brief Title: Assessment of MDD Management in Andalusia
Acronym: PismaEP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NES-XXX-2011/3; PismaEP
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: MDD Management Strategies
Keywords: MDD, management, Andalusia, Database, PismaEP

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The main objectives of this study are to describe medical professionals responsible of the management of patients with MDD in a representative region of Andalusia (in terms of type of sites managing the disease, and referral to SC criteria); Describe MDD patient characteristics at inclusion in the PISMA-Ep Study; and to evaluate those factors associated to a higher incidence of referral from PC to SC.

DETAILED DESCRIPTION:
Assessment of MDD management strategies in Andalusia: A Sub-analysis of the PismaEP Study

ELIGIBILITY:
Inclusion Criteria:

* MDD Diagnosis Participants of the PismaEP study 18 yo. or older

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDD patients treated in Primary Care or Secondary Care in the Region of Granada and recruited for the PISMA-Ep Study
Sampling Method: Probability Sample
Enrollment: 5309 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Visits to Primary Care | From Jan 2010 to Jan 2011
Number of Visits to Secondary Care | From Jan 2010 to Jan 2011
Number of Referrals | From Jan 2010 to Jan 2011

SECONDARY OUTCOMES:
Demographics | From Jan 2010 to Jan 2011
Type of site | From Jan 2010 to Jan 2011
Type of therapeutic strategy | From Jan 2010 to Jan 2011
Type of disease | From Jan 2010 to Jan 2011
Severity of disease | From Jan 2010 to Jan 2011

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cervilla, MD, Principal Investigator — Hospital San Cecilio
Locations (1):
- Research Site, Granada, Spain

REFERENCES:
- See also: NIS-NES-XXX-2011-3 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=924&filename=NIS-NES-XXX-2011-3_Clinical_Study_Report_Synopsis.pdf